CLINICAL TRIAL: NCT04649827
Title: SARS-CoV-2 Epidemiology Study at e Referenced Hospital in Fortaleza, Brazil: ResCOVID Study
Brief Title: A Clinical Trial for Hospitalized Patients With COVID-19 in Ceará: ResCOVID Study
Acronym: ResCOVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Escola de Saúde Pública do Ceará (Other Government)
Responsible Party: Principal Investigator, Marcelo Alcantara Holanda, Director, Escola de Saúde Pública do Ceará
Other Study IDs: 3.948.100
Record Dates: First submitted 2020-11-26; First posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: COVID-19
Keywords: COVID-19; Hospitalization; Public Health
MeSH Terms: conditions — COVID-19 | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19: Patients with confirmed COVID-19 by RT-PCR or serological test
  Interventions: Other: Clinical Observation

INTERVENTIONS:
Other: Clinical Observation — This is an observational study, so there are no interventions. Investigators will collect data about demographics, comorbidities, medications, and other risk factors such as the severity of disease at admission, need for advanced life support, need for invasive mechanical ventilation and main outcomes during hospitalization.

SUMMARY:
This is a case series of patients with COVID-19 admitted to the northeast Brazil region, in a referenced hospital for COVID-19, during the 2020 COVID-19 pandemic. Data will be collected prospectively and retrospectively.

The main objective is to describe the characteristics of critically ill patients with COVID-19 and their clinical outcomes, and to identify risk factors associated with survival, to guide the strategy to mitigate the epidemic, both within each hospital and ICU and in public health management.

DETAILED DESCRIPTION:
The world's population has been recently dealing with a new infectious disease, SARS-CoV-2 epidemic, which was first reported in December 2019 in Wuhan, China. The virus transmission was rapidly spread around the globe and the World Health Organization declared it as a public health emergency and it has been reported that SARS-CoV-2 is related to high morbidity and mortality rates.

The total number of infected patients has risen fastly and at the end of February 2020, the first case in Brazil was confirmed, suggesting that the SARS-CoV-2 is a pandemic situation.

The clinical aspect of SARS-CoV-2 ranges from pneumonia to critically ill cases, including clinical treatment, mechanical ventilation, and SARS.

The acute respiratory failure of critically ill patients with COVID-19 has different aspects, including hypoxemia of difficult treatment, associated in some cases with clotting disorders, changes in immunity and inflammatory phenomena that pose challenges for the management of these patients, whose mortality can be higher than expected.

The Public Health School in Fortaleza, Ceara, Brazil, implemented an action plan that provides several actions against COVID-19, including a specialized hospital and crew to treat these patients. Knowing the characteristics of critically ill patients with COVID-19 and their clinical outcomes is extremely important to inform clinical decision-making and to guide the strategy to mitigate the epidemic, both within each hospital and ICU and in public health management.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed COVID-19

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed COVID-19 by RT-PCR or sorological test, who are admitted at the referenced hospital in Fortaleza, Brazil.
  Data will be collected prospectively for patients admitted to the ICU after the date of study approval and retrospectively for patients admitted to the ICU during the COVID-19 epidemic in Fortaleza, but before the study was initiated.
  A sample size of 1000 patients was initially anticipated. As the epidemic in Fortaleza grew fast and it is one of the most affected regions in Brazil. The present study has no risks for participants since there are no new therapy or treatment to be tested. The investigators intend to collect data about all patients with COVID-19 admitted into the Hospital and at the ICU during the study period, possibly more than the anticipated sample size.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-04-02 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
ICU outcome | up to 60 days
  the proportion of patients who survive to ICU discharge

SECONDARY OUTCOMES:
Hospital outcome | up to 90 days
  the proportion of patients who survive to hospitalization
Mechanical ventilation | up to 60 days
  Mechanical ventilation time
Hospital complications | up to 90 days
  percentage of patients who developed complications during the hospitalization, both at ICU and during total hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo A Holanda, PHD, Principal Investigator — Escola Saude Publica
Locations (1):
- Hospital Leonardo Da Vinci, Fortaleza, Ceará, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
The investigators haven't developed a plan for sharing, but would be open to share unidentified data for research or public health purposes